CLINICAL TRIAL: NCT00845273
Title: Special Investigation For Long-term Use Of Macugen (Regulatory Post Marketing Commitment Plan).
Brief Title: Long-Term Use Of Pegaptanib In Patients For Subfoveal Choroidal Neovascularization Secondary To Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5751033
Record Dates: First submitted 2008-12-09; First posted 2009-02-18 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Macular Degeneration
Keywords: Subfoveal choroidal neovascularization secondary to age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pegaptanib sodium: Patients administered Pegaptanib sodium.
  Interventions: Drug: Pegaptanib sodium

INTERVENTIONS:
Drug: Pegaptanib sodium — Macugen Intravitreous Injection Kit 0.3mg depending on the Investigator prescription.
  Frequency and duration are according to Package Insert as follows. "Pegaptanib sodium is administered intravitreously once every 6 weeks at a dose level of 0.3 mg (on an oligonucleotide of pegaptanib basis )".
  Other Names: Macugen

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3) factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Macugen® should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Macugen® in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Macugen®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A5751033 prescribes the Macugen®).
Sampling Method: Probability Sample
Enrollment: 3538 (Actual)
Dates: Start 2008-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Factors considered to affect the safety and/or efficacy of this drug. | 2 years
The incidence of adverse drug reactions in this surveillance. | 2 years
Adverse drug reaction not expected from the LPD (unknown adverse drug reaction). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer